CLINICAL TRIAL: NCT02948855
Title: Study on Regulation of LncRNA to Regulatory B Cells(Bregs) Through Notch Pathway in Patients With Thymoma and Autoimmune Diseases
Brief Title: Regulation of LncRNA For Breg in Patients With Thymoma and Autoimmune Diseases
Status: Withdrawn | Type: Observational
Why Stopped: Improper design of the trial and no participants enrolled.
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: bc2016031
Record Dates: First submitted 2016-10-09; First posted 2016-10-31 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2016-10

CONDITIONS: Thymoma; Autoimmune Disease
Keywords: Long non-coding RNA（LncRNA）; Thymoma; Autoimmune disease; Notch2 Signaling pathway; Regulatory B cell（Breg）
MeSH Terms: conditions — Thymoma; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The patients of Thymoma complicated with autoimmune diseases:
  Thymoma tissues Lymph glands Peripheral blood Thymoma tissues and Lymph glands will be retained formalin and -80℃ refrigerator.
  Peripheral blood will be detected by flow cytometry.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Tm group: Simple thymoma group：The patients have suffered thymoma only and have no other complications.
- Tm+MG group: Thymoma complicated with myasthenia gravis (MG) group: The patients have suffered thymoma and myasthenia gravis in the mean time.
- Tm+MG+AD group: Thymoma complicated with myasthenia gravis and other autoimmune diseases (AD) group:
  The patients have suffered thymoma, myasthenia gravis and other autoimmune diseases in the mean time.

SUMMARY:
Initially investigators will find LncRNA which to be able to affect Notch2 signaling pathway; then confirm the relationship between Notch2 and LncRNA, and analysis the regulation mode of LncRNA to Notch2 signaling pathway, and to observe the correlation between LncRNA and thymoma complicated with autoimmune diseases.

DETAILED DESCRIPTION:
1. This study plans to research the correlation between Bregs and thymoma complicated with autoimmune diseases and the regulation the severity of the disease.
2. Clarify different expression levels of Notch2 signaling pathway in thymoma complicated with autoimmune diseases, and the effect on Regulatory B Cells(Bregs).
3. Find the effective regulation mode of Notch2 signaling pathway and the regulation of Bregs cell development and function in LncRNA.

ELIGIBILITY:
Inclusion Criteria:

* (1) The patients with the diagnosis of mediastinal tumors (thymoma, thymic hyperplasia);

  (2) The patients with the diagnosis of autoimmune diseases;

  (3) Age of 18 years or older which expected to stay in ICU for≥5 days.

  (4) APACHE II score > 15;

  (5) The patients or authorized clients agree to participate in the clinical trial and sign the informed consent.

Exclusion Criteria:

* (1) the patients with circulatory, respiratory failure and major organ dysfunction after being endangered and transferred to ICU;

  (2) patients with severe liver and renal dysfunction;

  (3) pregnant or lactating women;

  (4) patients who have not signed the informed consent;

  (5) any factors that may be expected to increase the risk of patients or other factors that may interfere with the outcome of clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. The patients with the diagnosis of mediastinal tumors (thymoma, thymic hyperplasia);
  2. The patients with the diagnosis of autoimmune diseases;
  3. Age of 18 years or older which expected to stay in ICU for≥5 days.
  4. APACHE II score > 15;
  5. The patients or authorized clients agree to participate in the clinical trial and sign the informed consent.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
The relationship between LncRNA and Notch2 signaling pathway | 2016.10.01~2018.09.31-up to 24 months
  Using of Real-Time Polymerase Chain Reaction(RT-PCR) and Western-Blot to find special LncRNA that can affect the Notch2 signaling pathway LncRNA's and Notch2 signaling pathway's gene and protein expression level Then, using of SiRNA to inhibit the expression of LncRNA or plasmid transfection to raise the expression of LncRNA, and observation of changes of Notch2 signaling pathway.

SECONDARY OUTCOMES:
The regulated effect of Notch2 signaling pathway to the development of Bregs and the cell function | 2016.10.01~2018.09.31-up to 24 months
  Peripheral blood was obtained from participants, and Regulatory B Cells(Bregs) were extracted and cultured.
  SiRNA-Notch2 to inhibit the expression of Notch2 signaling pathway and plasmid transfection of Notch2 to raise the expression of Notch2 signaling pathway, Then, observation of the quantity (*10^6/ml) and morphological changes of Bregs; the expression differences of Notch2 signaling pathway and content level (pg/ml) of Interleukin-10 (IL-10) in culture supernatant

OTHER OUTCOMES:
The relevance of Bregs and thymoma with autoimmune diseases | 2016.10.01~2018.09.31-up to 24 months
  Natural disease course (number of days) Treatment options: hormone dosage (mg), cytotoxic drug dosage (mg), 28 day mortality (%), treatment success rate.
  Laboratory examination: white blood cell (*10^9/L), hemoglobin (g/L), urinary protein (mg/L), titers of autoimmune antibody.
  Vital signs: heart rate (bpm), body temperature.

CONTACTS AND LOCATIONS:
Overall Officials: Donghao Wang, director, Study Director — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Strobel P, Hartmann E, Rosenwald A, Kalla J, Ott G, Friedel G, Schalke B, Kasahara M, Tomaru U, Marx A. Corticomedullary differentiation and maturational arrest in thymomas. Histopathology. 2014 Mar;64(4):557-66. doi: 10.1111/his.12279. Epub 2013 Nov 18. PMID 24236644
- [Background] Kessel A, Haj T, Peri R, Snir A, Melamed D, Sabo E, Toubi E. Human CD19(+)CD25(high) B regulatory cells suppress proliferation of CD4(+) T cells and enhance Foxp3 and CTLA-4 expression in T-regulatory cells. Autoimmun Rev. 2012 Jul;11(9):670-7. doi: 10.1016/j.autrev.2011.11.018. Epub 2011 Dec 2. PMID 22155204
- [Background] Klinker MW, Lundy SK. Multiple mechanisms of immune suppression by B lymphocytes. Mol Med. 2012 Feb 10;18(1):123-37. doi: 10.2119/molmed.2011.00333. PMID 22033729
- [Background] Bray SJ. Notch signalling: a simple pathway becomes complex. Nat Rev Mol Cell Biol. 2006 Sep;7(9):678-89. doi: 10.1038/nrm2009. PMID 16921404
- [Background] Matsumoto M, Baba A, Yokota T, Nishikawa H, Ohkawa Y, Kayama H, Kallies A, Nutt SL, Sakaguchi S, Takeda K, Kurosaki T, Baba Y. Interleukin-10-producing plasmablasts exert regulatory function in autoimmune inflammation. Immunity. 2014 Dec 18;41(6):1040-51. doi: 10.1016/j.immuni.2014.10.016. Epub 2014 Nov 4. PMID 25484301
- [Background] Mauri C, Menon M. The expanding family of regulatory B cells. Int Immunol. 2015 Oct;27(10):479-86. doi: 10.1093/intimm/dxv038. Epub 2015 Jun 12. PMID 26071023